CLINICAL TRIAL: NCT04929548
Title: Exploratory Study of Triple-targeted Neoadjuvant Treatment of HER2-positive Breast Cancer With Pyrotinib in Combination With Trastuzumab and Pertuzumab
Brief Title: Exploratory Study of Neoadjuvant Treatment of HER2-positive Breast Cancer With Py in Combination With HP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Ph D, MD, Director, Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WuhanU
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant; Targeted Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECPy-THP Programs (Experimental): Epirubicin 100 mg/m2, iv cyclophosphamide 600 mg/m2, iv + Pyrotinib 400 mg/d, po 4-week treatment, sequential docetaxel 80 mg/m2, iv + trastuzumab 6 mg/kg (first dose 8 mg/kg), iv + patuximab 420 mg (first dose 840 mg), iv ,po 4 weeks of treatment
  Interventions: Drug: Pyrotinib Maleate Tablets

INTERVENTIONS:
Drug: Pyrotinib Maleate Tablets — Addition of Pyrotinib in the EC phase to the standard treatment EC-THP regimen recommended by the guidelines.

SUMMARY:
This study is a single-arm, single-center exploratory clinical study. Twenty patients with early-stage HER2-positive breast cancer are planned to be included, and the primary objective is to evaluate the efficacy of neoadjuvant regimen of Pyrotinib in combination with trastuzumab + pertuzumab.

DETAILED DESCRIPTION:
Recruiting patients with clinical stage II to III HER2-positive breast cancer for primary treatment, eligible subjects will be enrolled as follows： This study is a single-arm, single-center exploratory clinical study. Twenty patients with early-stage HER2-positive breast cancer are planned to be included, and the primary objective is to evaluate the efficacy of neoadjuvant regimen of Pyrotinib in combination with trastuzumab + pertuzumab.Eligible subjects who met the enrollment criteria and signed the informed consent form entered the trial period and received epirubicin 100 mg/m2, iv cyclophosphamide 600 mg/m2, iv + Pyrotinib 400 mg/d, po for 4 weeks, sequential docetaxel 80 mg/m2, iv + trastuzumab 6 mg/kg (first dose 8 mg/kg), iv + pertuzumab 420 mg (first dose 840 mg), iv ,po 4 cycles of treatment. Surgery was performed at the end of the above treatment cycles, and adjuvant targeted therapy was continued after surgery: trastuzumab + patuximab for 1 year.

Eligible subjects (20) who met the nadir criteria and signed the informed consent form entered the trial period and received the ECPy-THP regimen: i.e., epirubicin 100 mg/m2, iv + cyclophosphamide 600 mg/m2, iv + Pyrotinib 400 mg/d, po 4 cycles, sequential docetaxel 80 mg/m2, iv + trastuzumab 6 mg/kg (first dose 8 mg/kg), iv + patuximab 420 mg (first dose 840 mg), iv, po 4 cycles of treatment. If the efficacy of 4 cycles was evaluated as PD or SD, the regimen was promptly adjusted for surgical treatment.

Surgery was performed at the end of the above treatment cycles, and adjuvant targeted therapy was continued after surgery: patients who reached pCR continued trastuzumab + pertuzumab for 1 year, and non-pCR patients were treated according to the guideline-recommended backline regimen.

All patients underwent surgery or radiotherapy continuation within 16-20 d after completion of the neoadjuvant chemotherapy cycle, and the efficacy was assessed 1 to 2 d before continuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-70 years.
* ECOG score must be 0 or 1.
* Patients with clinical stage II to III new breast cancer, all diagnosed by hollow-core needle aspiration biopsy pathological histology prior to treatment and surgically resectable breast cancer with positive immunohistochemical staining (IHC) for HER2 (3+) or HER2 (2+) supplemented with fluorescence in situ hybridization technique (FISH).
* The presence of at least one measurable lesion according to RECIST 1.1 criteria.
* Exclusion of distant metastases by abdominal B-ultrasound, chest X-ray and whole-body bone scan prior to neoadjuvant chemotherapy, and for lymph nodes in the enlarged area fine needle aspiration cytology is required to clarify the presence of tumor metastases without a history of remaining malignancies.
* Expected survival of not less than 12 weeks.
* No previous treatment, including chemotherapy, radiotherapy, targeted therapy, and biologic therapy. -Exclusion Criteria

Exclusion Criteria:

* Female patients of childbearing age who are pregnant, breastfeeding, or unwilling to use effective contraception throughout the trial period.
* Patients with combined severe cardiac, hepatic, renal, or endocrine system diseases and with expected survival of < 2 years for the above diseases.
* Inability to swallow, intestinal obstruction, the presence of other factors affecting drug administration and absorption or a history of allergy to this drug
* Karnofsky scale score below 60
* Patients with metastatic breast cancer or bilateral breast cancer.
* Patients with inflammatory breast cancer.
* Those with a left ventricular ejection fraction (LVEF) <55% on echocardiography
* Those who are deemed by the personnel to be otherwise unsuitable for clinical trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-05 (Estimated); Primary Completion 2022-01-05 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 6 months
  Complete remission of pathology

SECONDARY OUTCOMES:
RFS | 5 years
  RELAPSE-FREE SURVIVAL
OS | 5 years
  Overall survival

IPD SHARING:
Plan to Share IPD: Undecided